CLINICAL TRIAL: NCT03315689
Title: A Randomized, Double-blind, Vehicle-controlled Multicenter Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of ATI-50002 Topical Solution Administered Twice-Daily for 28 Days in Adult Subjects With Alopecia Universalis and Alopecia Totalis With a 12-Month Long-Term Open-Label Extension
Brief Title: Safety and Pharmacokinetic Study of ATI-50002 in Subjects With Alopecia Universalis (AU) and Alopecia Totalis (AT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATI-50002-AA-202
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Results first posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Alopecia Universalis (AU); Alopecia Totalis (AT)
MeSH Terms: conditions — Alopecia universalis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vehicle (Placebo Comparator): Vehicle
  Interventions: Drug: Vehicle
- Active (Experimental): ATI-50002 Topical Solution
  Interventions: Drug: ATI-50002

INTERVENTIONS:
Drug: Vehicle — Vehicle Topical Solution
  Arms: Vehicle
Drug: ATI-50002 — ATI-50002 Topical Solution
  Arms: Active

SUMMARY:
The primary objective is to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of ATI-50002 Topical Solution compared to vehicle in subjects with AU and AT.

DETAILED DESCRIPTION:
This study is designed to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of ATI-50002 Topical Solution in patients with Alopecia Universalis and Alopecia Totalis. Concentrations of ATI-50002 in the blood and skin will be assessed after 28 days of treatment with ATI-50002 Topical Solution.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and willing to sign an Informed Consent Form (ICF).
* Male or non-pregnant, non-nursing female ≥18 years old at the time of informed consent.
* Have a clinical diagnosis of stable, clinically typical, AU or AT.
* Have a duration of the current episode of AU or AT for a minimum of 6 months and a maximum of seven years.
* Be willing and able to follow all study instructions and to attend all study visits.

Exclusion Criteria:

* Females who are nursing, pregnant, or planning to become pregnant for the duration of the study including 30 days after the last application of study medication.
* Patchy alopecia areata, diffuse alopecia areata or a history of an atypical pattern of Alopecia Areata (AA) (e.g., ophiasis, sisaihpo).
* Active skin disease on the scalp (such as psoriasis or seborrheic dermatitis) or a history of skin disease on the scalp that in the opinion of the investigator would interfere with the study assessments of efficacy or safety.
* Active scalp trauma or other condition affecting the scalp that, in the investigator's opinion, may affect the course of AU or AT or interfere with the study conduct or evaluations.
* The presence of a permanent or difficult to remove hairpiece or wig that will, in the opinion of the investigator, interfere with study assessments if not removed at each visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Aclaris Investigational Site, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Vehicle Topical Solution: Vehicle Topical Solution applied twice daily.
- ATI-50002 0.46% Topical Solution: ATI-50002 0.46% Topical Solution applied twice daily.
Period: Double-blind Period = 28 Days
Arm/Group | Vehicle Topical Solution | ATI-50002 0.46% Topical Solution
Started | 4 | 7
Completed | 3 | 7
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Open Label Extension = 52 Weeks
Arm/Group | Vehicle Topical Solution | ATI-50002 0.46% Topical Solution
Started (All participants entering the Open Label Extension were provided ATI-50002 0.46% Topical Solution.) | 0 | 10
Completed | 0 | 7
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle Topical Solution | ATI-50002 0.46% Topical Solution | Total
Number analyzed (Participants) | 4 | 7 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 8
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 4 | 6
  Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 7 | 11
Fitzpatrick Skin Type [Count of Participants; unit: Participants]
  I - Always Burns | 0 | 2 | 2
  II - Burns Easily | 3 | 2 | 5
  III - Burns Moderately | 0 | 0 | 0
  IV - Burns Minimally | 0 | 1 | 1
  V - Rarely Burns | 1 | 2 | 3
  VI - Never Burns | 0 | 0 | 0
Current Clinical Type of Alopecia [Count of Participants; unit: Participants]
  Totalis | 1 | 3 | 4
  Universalis | 3 | 4 | 7
Time Since Onset of Current Episode of AU or AT [Mean (Standard Deviation); unit: Weeks] | 145.8 (128.58) | 218.3 (122.10) | 191.9 (123.47)

OUTCOME MEASURES:

1. Primary Outcome: Double Blind Period: ATI-50002 Levels in Scalp Biopsy (ng/g) - Pharmacodynamic (PD) Population at Day 2 and Day 29
Description: ATI-50002 levels in scalp biopsies taken at Visits 3 (Day 2) and 7 (Day 29).
Time Frame: Day 2 - Day 29
Population: All randomized patients who have a valid assessment at baseline and the subsequent timepoint being reported are included.
Measure: Mean (Standard Deviation); unit: ng/g
Arm/Group | Vehicle | Active
Number analyzed (Participants) | 3 | 6
ng/g
  V3 - Day 2 | 166.0 (83.44) | 579.7 (322.36)
  V7 - Day 29 | NA (NA) — Of the 3 participants with available samples for analysis, all results were below quantifiable limits where the lower limit of quantification was 100 ng/g. | 5710.0 (3647.87)

2. Secondary Outcome: Open Label Extension: Mean Change From Baseline in the Severity of Alopecia Tool (SALT) Score at Week 52
Description: The Severity of Alopecia Tool (SALT) score is a physician administered scale measuring the amount of scalp without any terminal hair. Possible scores range from 0 (no scalp hair loss) to 100 (complete scalp hair loss). A negative change in the SALT score over time represents hair regrowth.
Time Frame: Baseline - Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- ATI-50002 0.46% Topical Solution OLE: ATI-50002 0.46% Topical Solution applied twice daily during the open label extension period of the study
Arm/Group | ATI-50002 0.46% Topical Solution OLE
Number analyzed (Participants) | 4
score on a scale | -15.0 (16.21)

3. Secondary Outcome: Open Label Extension: Mean Change From Baseline in the Severity of Alopecia Tool (SALT) Score at Week 40
Description: as for outcome 2
Time Frame: Baseline - Week 40
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution OLE
Number analyzed (Participants) | 4
score on a scale | -8.8 (12.84)

4. Secondary Outcome: Open Label Extension: Mean Change From Baseline in the Severity of Alopecia Tool (SALT) Score at Week 28
Description: as for outcome 2
Time Frame: Baseline - Week 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution OLE
Number analyzed (Participants) | 8
score on a scale | -6.1 (11.91)

5. Secondary Outcome: Open Label Extension: Change From Baseline in Alopecia Density and Extent Score (ALODEX) at Week 28
Description: The Alopecia Density and Extent (ALODEX) score is a measurement of the amount of scalp with terminal hair loss assessed by the investigator. ALODEX breaks the scalp up into a grid of 1% scalp surface areas and assigns density rating in each area on a 10 point scale of hair loss (0= no hair loss to 10 = complete baldness). Summation of scores from each 1% scalp surface area provides an overall score which may range from 0 (no scalp hair loss) to 100 (complete baldness). A negative change in the ALODEX score over time represents hair regrowth.
Time Frame: Baseline - Week 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution OLE
Number analyzed (Participants) | 8
score on a scale | -7.1 (12.71)

6. Secondary Outcome: Open Label Extension: Change From Baseline in Alopecia Density and Extent Score (ALODEX) at Week 40
Description: as for outcome 5
Time Frame: Baseline - Week 40
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution OLE
Number analyzed (Participants) | 4
score on a scale | -9.5 (10.66)

7. Secondary Outcome: Open Label Extension: Change From Baseline in Alopecia Density and Extent Score (ALODEX) at Week 52
Description: as for outcome 5
Time Frame: Baseline - Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution OLE
Number analyzed (Participants) | 4
score on a scale | -12.0 (11.58)

8. Secondary Outcome: Open Label Extension: Mean Change in Subject's Eyebrow Assessment (SEA) at Week 28
Description: The Subject Eyebrow Assessment (SEA) is the subject's assessment of the appearance of eyebrow hair present on the affected eyebrow(s) at a particular point in time. The SEA is a five-point VRS ranging from "0 - No eyebrow hair", "1 - A little eyebrow hair", "2 - Some eyebrow hair", "3 - Most eyebrow hair", and "4 - Full eyebrow hair" with a recall period of "right now". A positive change over time represents eyebrow regrowth (better outcome).
Time Frame: Week 4 - Week 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution OLE
Number analyzed (Participants) | 8
score on a scale | 0.4 (0.90)

9. Secondary Outcome: Open Label Extension: Mean Change in Subject's Eyebrow Assessment (SEA) at Week 40
Description: as for outcome 8
Time Frame: Week 4 - Week 40
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution OLE
Number analyzed (Participants) | 4
score on a scale | 0.5 (1.58)

10. Secondary Outcome: Open Label Extension: Mean Change in Subject's Eyebrow Assessment (SEA) at Week 52
Description: as for outcome 8
Time Frame: Week 4 - Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution OLE
Number analyzed (Participants) | 4
score on a scale | 0.6 (1.38)

11. Secondary Outcome: Open Label Extension: Mean Change in Clinician's Eyebrow Assessment (CEA) at Week 28
Description: The Clinician's Eyebrow Assessment (CEA) is the investigator's assessment of the appearance of eyebrow hair present on the affected eyebrow(s) at a particular point in time. The CEA is a five-point VRS ranging from "0 - No eyebrow hair", "1 - A little eyebrow hair", "2 - Some eyebrow hair", "3 - Most eyebrow hair", and "4 - Full eyebrow hair" with a recall period of "right now". A positive change over time represents eyebrow regrowth (better outcome).
Time Frame: Week 4 - Week 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution OLE
Number analyzed (Participants) | 8
score on a scale | 0.1 (1.16)

12. Secondary Outcome: Open Label Extension: Mean Change in Clinician's Eyebrow Assessment (CEA) at Week 40
Description: as for outcome 11
Time Frame: Week 4 - Week 40
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution OLE
Number analyzed (Participants) | 4
score on a scale | 0.6 (1.11)

13. Secondary Outcome: Open Label Extension: Mean Change in Clinician's Eyebrow Assessment (CEA) at Week 52
Description: as for outcome 11
Time Frame: Week 4 - Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-50002 0.46% Topical Solution OLE
Number analyzed (Participants) | 4
score on a scale | 0.8 (1.19)

14. Secondary Outcome: Open Label Extension: Subject Global Impression of Treatment Satisfaction (SGIS) Week 28
Description: The Subject Global Impression of Treatment Satisfaction (SGIS) is a 7-point descriptive scale with a recall period of "right now". The SGIS was completed by subjects during the Open Label period of the study. Scale response options ranged from "1: Extremely Satisfied", "2: Moderately Satisfied", "3: A little Satisfied", "4: Neither Satisfied or Dissatisfied", "5: A little Dissatisfied", "6: Moderately Dissatisfied", or "7: Extremely Dissatisfied" and are used to capture how satisfied or dissatisfied subjects are with the study medication treatment received for their alopecia areata.
Time Frame: Week 28
Population: All patients who have a valid assessment at the timepoint being reported are included.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-50002 0.46% Topical Solution OLE
Number analyzed (Participants) | 8
Participants
  1: Extremely Satisfied | 0
  2: Moderately Satisfied | 2
  3: A little Satisfied | 1
  4: Neither Satisfied or Dissatisfied | 1
  5: A little Dissatisfied | 0
  6: Moderately Dissatisfied | 1
  7: Extremely Dissatisfied | 3

15. Secondary Outcome: Open Label Extension: Subject Global Impression of Treatment Satisfaction (SGIS) Week 40
Description: as for outcome 14
Time Frame: Week 40
Population: All patients who have a valid assessment at the timepoint being reported are included.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-50002 0.46% Topical Solution OLE
Number analyzed (Participants) | 4
Participants
  1: Extremely Satisfied | 0
  2: Moderately Satisfied | 2
  3: A little Satisfied | 0
  4: Neither Satisfied or Dissatisfied | 1
  5: A little Dissatisfied | 0
  6: Moderately Dissatisfied | 0
  7: Extremely Dissatisfied | 1

16. Secondary Outcome: Open Label Extension: Subject Global Impression of Treatment Satisfaction (SGIS) Week 52
Description: as for outcome 14
Time Frame: Week 52
Population: All patients who have a valid assessment at the timepoint being reported are included.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-50002 0.46% Topical Solution OLE
Number analyzed (Participants) | 4
Participants
  1: Extremely Satisfied | 0
  2: Moderately Satisfied | 2
  3: A little Satisfied | 0
  4: Neither Satisfied or Dissatisfied | 1
  5: A little Dissatisfied | 0
  6: Moderately Dissatisfied | 0
  7: Extremely Dissatisfied | 1

17. Secondary Outcome: Open Label Extension: Severity of Alopecia Tool (SALT) Scores, Relative Percent Regrowth (%) at Week 24 From Baseline
Description: The Severity of Alopecia Tool (SALT) score is a physician administered scale measuring the amount of scalp without any terminal hair assessed by the investigator. A positive percent change over time represents hair regrowth (better outcome).
Time Frame: Baseline - Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ATI-50002 0.46% Topical Solution OLE
Number analyzed (Participants) | 8
percent change | 6.3 (12.14)

18. Secondary Outcome: Open Label Extension: Severity of Alopecia Tool (SALT Scores), Relative Percent Regrowth (%) at Week 40 From Baseline
Description: as for outcome 17
Time Frame: Baseline - Week 40
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ATI-50002 0.46% Topical Solution OLE
Number analyzed (Participants) | 4
percent change | 9.0 (13.01)

19. Secondary Outcome: Open Label Extension: The Severity of Alopecia Tool (SALT) Scores, Relative Percent Regrowth (%) at Week 52 From Baseline
Description: as for outcome 17
Time Frame: Baseline - Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ATI-50002 0.46% Topical Solution OLE
Number analyzed (Participants) | 4
percent change | 15.5 (16.77)

20. Secondary Outcome: Open Label Extension: The Alopecia Density and Extent (ALODEX) Scores, Relative Percent Regrowth (%) at 24 Weeks
Description: The Alopecia Density and Extent (ALODEX) score is a measurement of the amount of scalp with terminal hair loss assessed by the investigator. ALODEX breaks the scalp up into a grid of 1% scalp surface areas and assigns density rating in each area on a 10 point scale of hair loss (0= no hair loss to 10 = complete baldness). Summation of scores from each 1% scalp surface area provides an overall score which may range from 0 (no scalp hair loss) to 100 (complete baldness). A positive percent change over time represents hair regrowth (better outcome).
Time Frame: Baseline - Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ATI-50002 0.46% Topical Solution OLE
Number analyzed (Participants) | 8
percent change | 7.2 (12.88)

21. Secondary Outcome: Open Label Extension: The Alopecia Density and Extent (ALODEX) Scores, Relative Percent Regrowth (%) at 40 Weeks
Description: The Alopecia Density and Extent (ALODEX) score is a measurement of the amount of scalp with terminal hair loss assessed by the investigator at Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24. ALODEX breaks the scalp up into a grid of 1% scalp surface areas and assigns density rating in each area on a 10 point scale of hair loss (0= no hair loss to 10 = complete baldness). Summation of scores from each 1% scalp surface area provides an overall score which may range from 0 (no scalp hair loss) to 100 (complete baldness). A positive percent change over time represents hair regrowth (better outcome).
Time Frame: Baseline - Week 40
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ATI-50002 0.46% Topical Solution OLE
Number analyzed (Participants) | 4
percent change | 9.6 (10.81)

22. Secondary Outcome: Open Label Extension: The Alopecia Density and Extent (ALODEX) Scores, Relative Percent Regrowth (%) at 52 Weeks
Description: as for outcome 20
Time Frame: Baseline - Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ATI-50002 0.46% Topical Solution OLE
Number analyzed (Participants) | 4
percent change | 12.2 (11.74)

ADVERSE EVENTS:
Time Frame: Double blind period = 28 days; Open label extension period = 12 months; Reporting of non-serious AEs started with each subject's first study medication application and continued until the end of the subject's last study visit. Reporting for SAEs started when the subject signed the informed consent document and continued until the end of the subject's last visit.
Groups:
- Vehicle Topical Solution: Vehicle Topical Solution applied twice daily during the double blind period of the study.
- ATI-50002 0.46% Topical Solution: ATI-50002 0.46% Topical Solution applied twice daily during the double blind period of the study
Arm/Group | Vehicle Topical Solution | ATI-50002 0.46% Topical Solution | ATI-50002 0.46% Topical Solution OLE
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/7 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/7 | 1/10
Other Adverse Events (participants affected / at risk) | 1/4 | 1/7 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Topical Solution (N=4) | ATI-50002 0.46% Topical Solution (N=7) | ATI-50002 0.46% Topical Solution OLE (N=10)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Topical Solution (N=4) | ATI-50002 0.46% Topical Solution (N=7) | ATI-50002 0.46% Topical Solution OLE (N=10)
Application site erosion (General disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-14): https://cdn.clinicaltrials.gov/large-docs/89/NCT03315689/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/89/NCT03315689/SAP_001.pdf